CLINICAL TRIAL: NCT02021123
Title: Pharmacokinetics of Anidulafungin (Ecalta ®) Given Intravenously as Prophylaxis to Obese Patients With Risk of Invasive Fungal Infection Undergoing Gastric Bypass Surgery.
Brief Title: Anidulafungin Pharmacokinetics Given as a Single Intravenous Dose to Obese Patients (ADOPT)
Acronym: ADOPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 13.06
Record Dates: First submitted 2013-11-29; First posted 2013-12-27 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Obesity Morbid
Keywords: Anidulafungin; Gastric bypass; Morbidly obese; Pharmacokinetics; Prophylaxis; Yeast infection
MeSH Terms: conditions — Obesity, Morbid | interventions — Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anidulafungin 100 mg single dose (Experimental): 100 mg single dose anidulafungin pre-surgery (gastric bypass)
  Interventions: Drug: Anidulafungin 100mg single dose iv

INTERVENTIONS:
Drug: Anidulafungin 100mg single dose iv — Anidulafungin 100mg single dose iv pre-surgery (gastric bypass)
  Other Names: Ecalta

SUMMARY:
Because anidulafungin is generally well tolerated and appears to have limited interaction with other drugs, it is a potential important agent in the treatment of invasive fungal infections. Although anidulafungin is approved for the treatment of invasive candidiasis in adult non-neutropenic patients, dosing guidelines for anidulafungin in (morbidly) obese patients are not available. Subsequently, the pharmacokinetic profile of anidulafungin (as well as other echinocandins) in this specific patient population is still largely unknown. During endoscopic gastric bypass surgery, patients are more prone to various kinds of infection, justifying the prophylactic use of anidulafungin in this specific cohort of patients.

To build a valid pharmacokinetic model, obese patients with a BMI ≥ 40 undergoing endoscopic gastric bypass surgery will receive a single dose of 100 mg anidulafungin (besides standard anti-bacterial prophylaxis) and a PK-curve will be drawn. These PK-values can then be compared to the pharmacokinetics in a normal-weight group.

DETAILED DESCRIPTION:
All obese patients with a BMI ≥ 40 kg/m2 undergoing endoscopic gastric bypass surgery who receive a prophylactic single dose of 100 mg anidulafungin will be included in the analysis. A PK curve will be determined after administration of anidulafungin at t=0.5, 1, end of infusion, 2, 4, 6, 8, 10, 12, 24, and 48 and (if feasible) 72 hours post infusion (n=12 samples). Blood samples (4 mL) on PK days will be taken to obtain at least 2.0 mL of plasma.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a BMI ≥40 kg/m2 and is undergoing endoscopic gastric bypass surgery.
2. Subject is at least 18 years of age on the day of screening.
3. If subject is female: neither pregnant, nor able to become pregnant and is not nursing an infant.
4. Subject or legal representatives are able and willing to sign the Informed Consent before screening evaluations.

Exclusion Criteria:

1. Documented history of sensitivity to medicinal products or excipients similar to those found in the echinocandin preparation.
2. History of, or current abuse of drugs, alcohol or solvents.
3. Inability to understand the nature of the trial and the procedures required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
anidulafungin area under the curve | 0-72 h after single dose
  The primary outcome measurement will be the area under the plasma concentration-time curve (AUC) from time 0 to infinitive (inf) post infusion (AUC0- inf) value of anidulafungin. This will be determined by use of the log-linear trapezoidal rule. Peak plasma concentrations (Cmax) will be directly observed from the data. The elimination rate constant will be determined by linear regression of the terminal points of the log-linear plasma concentration time curve. Clearance (CL) will be calculated as dose/AUC0- inf.

SECONDARY OUTCOMES:
Predict long-term exposure after repeated dosing by using a pharmacokinetic model of anidulafunign in obese patients by using AUC(0-inf), Cmax, elimination half-life and clearance. | PK curve on day 1-3
  Simulate pharmacokinetics of anidulafungin after obtaining all plasma concentrations using modeling software to predict long-term exposure. For this, area under the plasma concentration-time curve (AUC) from time 0 to infinitive (inf) post infusion (AUC0- inf), peak plasma concentration (Cmax), elimination half-life and clearance values of anidulafungin will be used (as calculated in outcome measure 1). The PK curve of day 1-3 will serve to calculate these values.

OTHER OUTCOMES:
adverse events | 0-72 h after dosing
  adverse events will be collected and reported

CONTACTS AND LOCATIONS:
Overall Officials: Roger JM Brüggemann, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - St. Antonius hospital, Nieuwegein

REFERENCES:
- [Result] Lempers VJ, van Rongen A, van Dongen EP, van Ramshorst B, Burger DM, Aarnoutse RE, Knibbe CA, Bruggemann RJ. Does Weight Impact Anidulafungin Pharmacokinetics? Clin Pharmacokinet. 2016 Oct;55(10):1289-1294. doi: 10.1007/s40262-016-0401-8. PMID 27142114